CLINICAL TRIAL: NCT00945750
Title: A Single-Dose, Open-Label, Three-Period Crossover Study to Assess the Bioequivalence of Famotidine 20 mg Film-Coated Tablets (FCT) Compared to Famotidine 20 mg Chewable Tablets (CT) Without Water and Famotidine 20 mg Chewable Tablets (CTw) With Water (Protocol 144)
Brief Title: A Study to Assess the Bioequivalence of Famotidine Chewable Tablets and Film-Coated Tablets (0208-144)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0208-144; 2009_621 (Other: Merck Registration Number)
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Heartburn
MeSH Terms: conditions — Heartburn | interventions — Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1: FCT with water → CT without water → CT with water (Experimental): Participants received famotidine 20 mg FCT as a single dose with 120 mL of water (Period 1), followed by a 5- to 7-day washout, followed by famotidine 20 mg CT as a single dose without water (Period 2), followed by a 5- to 7-day washout, followed by famotidine 20 mg CT as a single dose with 120 mL of water (Period 3).
  Interventions: Drug: Famotidine FCT; Drug: Famotidine CT
- Sequence 2: CT without water → CT with water → FCT with water (Experimental): Participants received famotidine 20 mg CT as a single dose without water (Period 1), followed by a 5- to 7-day washout, followed by famotidine 20 mg CT as a single dose with 120 mL of water (Period 2), followed by a 5- to 7-day washout, followed by famotidine 20 mg FCT as a single dose with 120 mL of water (Period 3).
  Interventions: Drug: Famotidine FCT; Drug: Famotidine CT
- Sequence 3: CT with water → FCT with water → CT without water (Experimental): Participants received famotidine 20 mg CT as a single dose with 120 mL of water (Period 1), followed by a 5- to 7-day washout, followed by famotidine 20 mg FCT as a single dose with 120 mL of water (Period 2), followed by a 5- to 7-day washout, followed by famotidine 20 mg CT as a single dose without water (Period 3).
  Interventions: Drug: Famotidine FCT; Drug: Famotidine CT
- Sequence 4: FCT with water → CT with water → CT without water (Experimental): Participants received famotidine 20 mg FCT as a single dose with 120 mL of water (Period 1), followed by a 5- to 7-day washout, followed by famotidine 20 mg as a single dose with 120 mL of water (Period 2), followed by a 5- to 7-day washout, followed by famotidine 20 mg CT as a single dose without water (Period 3).
  Interventions: Drug: Famotidine FCT; Drug: Famotidine CT
- Sequence 5: CT without water → FCT with water → CT with water (Experimental): Participants received famotidine 20 mg CT as a single dose without water (Period 1), followed by a 5- to 7-day washout, followed by famotidine 20 mg FCT as a single dose with 120 mL of water (Period 2), followed by a 5- to 7-day washout, followed by famotidine 20 mg CT as a single dose with 120 mL of water (Period 3).
  Interventions: Drug: Famotidine FCT; Drug: Famotidine CT
- Sequence 6: CT with water → CT without water → FCT with water (Experimental): Participants received famotidine 20 mg CT as a single dose with 120 mL of water (Period 1), followed by a 5- to 7-day washout, followed by famotidine 20 mg CT as a single dose without water (Period 2), followed by a 5- to 7-day washout, followed by famotidine 20 mg FCT as a single dose with 120 mL of water (Period 3).
  Interventions: Drug: Famotidine FCT; Drug: Famotidine CT

INTERVENTIONS:
Drug: Famotidine FCT — Famotidine 20 mg oral film-coated tablet taken once daily
Drug: Famotidine CT — Famotidine 20 mg oral chewable tablet taken once daily

SUMMARY:
This study will determine whether the CT formulation of famotidine taken with and without water is bioequivalent to the FCT formulation. The primary hypothesis is that the area under the concentration-time curve (AUC) and the maximum plasma concentration (Cmax) of a single dose of famotidine 20 mg CT without water are equivalent to a single dose of famotidine 20 mg FCT with water.

ELIGIBILITY:
Inclusion Criteria:

* Female participant is not pregnant or lactating
* Female of childbearing potential must use reliable means of contraception during the course of the study
* Is in good health
* Is able to abstain from smoking during the 24-hour periods before and during each treatment day

Exclusion Criteria:

* Has any major systemic disorders
* Has a history of ulcers, other Gastrointestinal (GI) disease, or GI surgery
* Has or has a history of any illness or condition that might interfere with optimal participation in the study
* Has a history of asthma or severe allergies to drugs or foods
* Currently uses prescribed or non-prescribed drugs on a regular basis
* Has a recent history of drug/alcohol abuse
* Consumes more than 6 cups of coffee per day
* Has unconventional or extreme dietary habits
* Has donated blood or has been in a clinical trial in which they received an investigational drug during the past 30 days
* Has a history of allergy or intolerance to antacids
* Is known to be pregnant or is not using reliable means of contraception

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2006-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0208-144&kw=0208-144&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to 1 of 6 treatment sequences of 1 of 3 treatments: (1) famotidine as a film-coated tablet (FCT) taken with water, (2) famotidine as a chewable tablet (CTw) taken with water, and (3) famotidine as a chewable tablet taken without water, over 3 study periods in a crossover design.
Groups:
- FCT With Water / CT Without Water / CT With Water: Participants received famotidine 20 mg FCT as a single dose with 120 mL of water, followed by a 5- to 7-day washout, followed by famotidine 20 mg CT as a single dose without water, followed by a 5- to 7-day washout, followed by famotidine 20 mg CT as a single dose with 120 mL of water.
- CT Without Water / CT With Water / FCT With Water: Participants received famotidine 20 mg CT as a single dose without water, followed by a 5- to 7-day washout, followed by famotidine 20 mg CT as a single dose with 120 mL of water, followed by a 5- to 7-day washout, followed by famotidine 20 mg FCT as a single dosewith 120 mL of water.
- CT With Water / FCT With Water / CT Without Water: Participants received famotidine 20 mg CT as a single dose with 120 mL of water, followed by a 5- to 7-day washout, followed by famotidine 20 mg FCT as a single dose with 120 mL of water, followed by a 5- to 7-day washout, followed by famotidine 20 mg CT as a single dose without water.
- FCT With Water / CT With Water / CT Without Water: Participants received famotidine 20 mg FCT as a single dose with 120 mL of water, followed by a 5- to 7-day washout, followed by famotidine 20 mg CT as a single dose with 120 mL of water, followed by a 5- to 7-day washout, followed by famotidine 20 mg CT as a single dose without water.
- CT Without Water / FCT With Water / CT With Water: Participants received famotidine 20 mg CT as a single dose without water, followed by a 5- to 7-day washout, followed by famotidine 20 mg FCT as a single dose with 120 mL of water, followed by a 5- to 7-day washout, followed by famotidine 20 mg CT as a single dose with 120 mL of water.
- CT With Water / CT Without Water / FCT With Water: Participants received famotidine 20 mg CT as a single dose with 120 mL of water, followed by a 5- to 7-day washout, followed by famotidine 20 mg CT as a single dose without water, followed by a 5- to 7-day washout, followed by famotidine 20 mg FCT as a single dose with 120 mL of water.
Period: Period I
Arm/Group | FCT With Water / CT Without Water / CT With Water | CT Without Water / CT With Water / FCT With Water | CT With Water / FCT With Water / CT Without Water | FCT With Water / CT With Water / CT Without Water | CT Without Water / FCT With Water / CT With Water | CT With Water / CT Without Water / FCT With Water
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period II
Arm/Group | FCT With Water / CT Without Water / CT With Water | CT Without Water / CT With Water / FCT With Water | CT With Water / FCT With Water / CT Without Water | FCT With Water / CT With Water / CT Without Water | CT Without Water / FCT With Water / CT With Water | CT With Water / CT Without Water / FCT With Water
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period III
Arm/Group | FCT With Water / CT Without Water / CT With Water | CT Without Water / CT With Water / FCT With Water | CT With Water / FCT With Water / CT Without Water | FCT With Water / CT With Water / CT Without Water | CT Without Water / FCT With Water / CT With Water | CT With Water / CT Without Water / FCT With Water
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FCT With Water / CT Without Water / CT With Water | CT Without Water / CT With Water / FCT With Water | CT With Water / FCT With Water / CT Without Water | FCT With Water / CT With Water / CT Without Water | CT Without Water / FCT With Water / CT With Water | CT With Water / CT Without Water / FCT With Water | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (5.32) [26 to 39] | 24.0 (7.38) [18 to 36] | 24.2 (4.38) [19 to 31] | 22.6 (3.51) [19 to 28] | 26.4 (6.11) [19 to 36] | 25.6 (6.50) [22 to 37] | 25.9 (6.09) [18 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 0 | 2 | 4 | 2 | 14
  Male | 1 | 3 | 5 | 3 | 1 | 3 | 16
Weight [Mean (Full Range); unit: Pounds] | 137.6 [106.9 to 158.4] | 163.0 [140.6 to 187.1] | 175.4 [139.6 to 195.0] | 147.9 [110.9 to 182.2] | 142.6 [113.9 to 185.1] | 180.4 [140.6 to 205.9] | 157.4 [106.9 to 205.9]

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From 0 to Infinity (AUC 0-∞) Following Single Dose Administration of Famotidine CT Without Water and Famotidine FCT With Water
Description: AUC values were natural log-transformed and analyzed using an analysis of variance (ANOVA) model. The ANOVA model contained factors for participant (random effect), period, treatment, and within-participant error.
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 24 hours post-dose
Population: Participants who completed the study
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL hr
Groups:
- Famotidine 20 mg CT Without Water: Famotidine 20 mg CT without water
- Famotidine 20 mg FCT With Water: Famotidine 20 mg FCT with 120 mL of water
Arm/Group | Famotidine 20 mg CT Without Water | Famotidine 20 mg FCT With Water
Number analyzed (Participants) | 30 | 30
ng/mL hr | 398.5 [350.9 to 452.6] | 394.8 [347.6 to 448.4]
Statistical Analysis 1: Comparison: Famotidine 20 mg CT Without Water vs Famotidine 20 mg FCT With Water; Test type: Non-Inferiority or Equivalence — If the 90% CI for the AUC geometric mean ratio (famotidine CT without water/famotidine FCT with water) is within the hypothesized interval (0.80 and 1.25), then the primary hypothesis of bioequivalence between CT without water and FCT with water is accepted; Geometric Mean Ratio = 1.01, 90% CI [0.94 to 1.09]

2. Primary Outcome: Peak Plasma Concentration (Cmax) of Famotidine Following Single Dose Administration of Famotidine CT Without Water and Famotidine FCT With Water
Description: Cmax values were natural log-transformed and analyzed using an ANOVA model. The ANOVA model contained factors for participant (random effect), period, treatment, and within-participant error.
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 24 hours post-dose
Population: Participants who completed the study
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Famotidine 20 mg CT Without Water | Famotidine 20 mg FCT With Water
Number analyzed (Participants) | 30 | 30
ng/mL | 67.2 [58.7 to 76.9] | 65.1 [56.9 to 74.5]
Statistical Analysis 1: Comparison: Famotidine 20 mg CT Without Water vs Famotidine 20 mg FCT With Water; Test type: Non-Inferiority or Equivalence — If the 90% CI for the Cmax geometric mean ratio (famotidine CT without water/famotidine FCT with water) is within the hypothesized interval (0.80 and 1.25), then the primary hypothesis of bioequivalence between CT without water and FCT with water is accepted; Geometric Mean Ratio = 1.03, 90% CI [0.93 to 1.14]

3. Secondary Outcome: AUC 0-∞ Following Single Dose Administration of Famotidine CT With Water and Famotidine FCT With Water
Description: AUC values were natural log-transformed and analyzed using an ANOVA model. The ANOVA model contained factors for participant (random effect), period, treatment, and within-participant error.
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 24 hours post-dose
Population: Participants who completed the study
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL hr
Groups:
- Famotidine 20 mg CT With Water: Famotidine 20 mg CT with 120 mL of water
Arm/Group | Famotidine 20 mg CT With Water | Famotidine 20 mg FCT With Water
Number analyzed (Participants) | 30 | 30
ng/mL hr | 440.1 [387.5 to 499.8] | 394.8 [347.6 to 448.4]
Statistical Analysis 1: Comparison: Famotidine 20 mg CT With Water vs Famotidine 20 mg FCT With Water; Test type: Superiority or Other; Geometric Mean Ratio = 1.11, 90% CI [1.04 to 1.20]

4. Secondary Outcome: Cmax of Famotidine Following Single Dose Administration of Famotidine CT With Water and Famotidine FCT With Water
Description: as for outcome 2
Time Frame: 0 (predose), 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 24 hours post-dose
Population: Participants who completed the study
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Famotidine 20 mg CT With Water | Famotidine 20 mg FCT With Water
Number analyzed (Participants) | 30 | 30
ng/mL | 73.0 [63.8 to 83.6] | 65.1 [56.9 to 74.5]
Statistical Analysis 1: Comparison: Famotidine 20 mg CT With Water vs Famotidine 20 mg FCT With Water; Test type: Superiority or Other; Geometric Mean Ratio = 1.12, 90% CI [1.02 to 1.24]

ADVERSE EVENTS:
Time Frame: Up to 31 days (including 14 day follow-up)
Groups:
- Famotidine 20 mg FCT With Water: Famotidine 20 mg FCT (film-coated tablet) with 120 mL of water
- Famotidine 20 mg CT Without Water: Famotidine 20 mg Chewable Tablet without water
- Famotidine 20 mg CT With Water: Famotidine 20 mg chewable tablet with 120 mL of water
Arm/Group | Famotidine 20 mg FCT With Water | Famotidine 20 mg CT Without Water | Famotidine 20 mg CT With Water
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 4/30 | 3/30 | 4/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Famotidine 20 mg FCT With Water (N=30) | Famotidine 20 mg CT Without Water (N=30) | Famotidine 20 mg CT With Water (N=30)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 3 (3) | 3 (4)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope vasovagal (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by Merck as confidential must be deleted prior to submission.